CLINICAL TRIAL: NCT00103792
Title: Comparative Study of the Efficacy of Induction Therapy With Cyclophosphamide or Mycophenolate Mofetil for Non-life-threatening Relapses of PR3- or MPO-ANCA Associated Vasculitis
Brief Title: Mycophenolate Mofetil for Treatment of Relapses of Wegener's Disease or Microscopic Polyangiitis (MPA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WG-MMF-1; UMCG-ANCA-MMF-1
Record Dates: First submitted 2005-02-14; First posted 2005-02-15 (Estimated); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Wegener's Granulomatosis; Vasculitis
Keywords: Induction therapy; ANCA-associated vasculitis; Wegener's granulomatosis; microscopic polyangiitis; mycophenolate mofetil; cyclophosphamide
MeSH Terms: conditions — Granulomatosis with Polyangiitis; Vasculitis; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Microscopic Polyangiitis | interventions — Mycophenolic Acid; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 MMF induction (Experimental): mycophenolate and steroids as remission induction, followed by azathioprine as maintenance therapy
  Interventions: Drug: mycophenolate mofetil
- 2 CYC induction (Active Comparator): cyclophosphamide and steroids, followed by maintenance therapy (azathioprine)
  Interventions: Drug: cyclophosphamide

INTERVENTIONS:
Drug: mycophenolate mofetil — 2000 mg mycophenolate mofetil per day combined with steroids for induction remission, followed by azathioprine standard maintenance therapy
  Arms: 1 MMF induction
Drug: cyclophosphamide — 2 mg/kg/d, combined with steroids, for remission induction, followed by standard azathioprine maintenance therapy
  Arms: 2 CYC induction

SUMMARY:
The purpose of this study is to determine the efficacy and safety of a new drug, mycophenolate mofetil, for the treatment of relapses of ANCA-associated vasculitis (Wegener's granulomatosis or microscopic polyangiitis). Therefore, we compare the standard therapy with cyclophosphamide to mycophenolate mofetil.

The investigators expect mycophenolate mofetil to be less toxic and almost equally effective as cyclophosphamide.

DETAILED DESCRIPTION:
Treatment of ANCA-associated vasculitis consists of two phases: remission induction with highly effective, but also relatively toxic drugs, and, secondly, after remission is achieved, maintenance therapy with less toxic drugs. The standard induction therapy of a relapse of Wegener's granulomatosis or microscopic polyangiitis consists of the combination of cyclophosphamide and prednisolone. Although this induction therapy is very effective, it is very toxic as well.

Searching for an alternative for cyclophosphamide, we will test the efficacy and safety of a new combination therapy with mycophenolate mofetil and prednisolone. We will compare the effect and safety of the standard induction therapy with the new therapy. When relapses occur, patients will be randomized for either the standard therapy with cyclophosphamide or for mycophenolate mofetil.

ELIGIBILITY:
Inclusion Criteria:

* First or second relapse ANCA-associated vasculitis
* PR3- or MPO-ANCA antibodies present or histological proof of relapse
* Adult

Exclusion Criteria:

* Severe alveolar bleeding or (imminent) respiratory failure
* Renal failure (serum creatinine >500 umol/L or dialysis)
* Maintenance therapy before start of study consisting of: cyclophosphamide > 100 mg/day or prednisolone >25 mg/day
* Intolerance or allergy for cyclophosphamide, mycophenolate mofetil or azathioprine
* Gravidity or inadequate anticonception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2004-12 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
remission induction rate | 6 months
disease free survival after 2 and 4 years | 2 and 4 years

SECONDARY OUTCOMES:
time to remission | 9 months
cumulative organ damage | 4 years
side-effects | 4 years
ANCA titres over time | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Coen Stegeman, MD PhD, Principal Investigator — UMCG Groningen
Locations (1):
- University Medical Centre Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Stegeman CA; Cohen Tervaert JW. Mycophenolate mofetil for remission induction in patients with active Wegener's Granulomatosis (WG) intolerant for cyclophosphamide. J Am Soc Nephrol(11):98A, 2000